CLINICAL TRIAL: NCT06808009
Title: Goal Directed Ammonia Lowering Therapy in Hyperammonemic ACLF Patients With no Overt HE to Reduce Major Adverse Liver Related Outcomes (GOAL Trial)- A Randomized Controlled Trial
Brief Title: Goal Directed Ammonia Lowering Therapy in Hyperammonemic ACLF Patients With no Overt HE to Reduce Major Adverse Liver Related Outcomes (GOAL Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-23
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Lactulose; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactulose and rifaximin (Experimental): T. Rifaximin 550 mg po bd Syp Lactulose to ensure 2-3 motions
  Interventions: Drug: Lactulose; Drug: Rifaximin
- Standard Medical Treatment (Active Comparator): Routine medicines, Albumin Iv antibiotics,Protein powder , branched chain amino acids
  Interventions: Other: Standard Medical treatment

INTERVENTIONS:
Drug: Lactulose — Syp lactulose
  Arms: lactulose and rifaximin
Drug: Rifaximin — Rifaximin
  Arms: lactulose and rifaximin
Other: Standard Medical treatment — Standard Medical treatment
  Arms: Standard Medical Treatment

SUMMARY:
SIRS in ACLF exacerbate adverse effects of ammonia - sarcopenia, infections, immune dysfunction, HE and organ dysfunction Persistent or incident hyperammonemia during first week of hospitalization in patients with ACLF is associated with increased risk of organ failure and death. Prospective studies on the efficacy of ammonia lowering therapies on major adverse liver related outcomes (MALO) (any of AARC III, bacterial infection, overt HE grade or death) in hyperammonemic ACLF patients with no overt HE are limited. In this study we aim to to compare the safety and efficacy of ammonia lowering therapy (goal directed lactulose and rifaximin) compared to SMT to prevent major liver related outcomes (MALO) (any of AARC III, bacterial infection, overt HE grade or death) in hyperammonemic ACLF patients with no overt HE.

DETAILED DESCRIPTION:
Hypothesis: Goal directed ammonia lowering therapy in hyperammonemic ACLF patients with no overt HE leads to reduced incidence of major adverse liver related outcomes (MALO) (any of AARC III, bacterial infection, overt HE grade or death) at day 7, 28 and day 90.

AIM:- To compare the safety and efficacy of ammonia lowering therapy (goal directed lactulose and rifaximin) compared to SMT to prevent major liver related outcomes (MALO) (any of AARC III, bacterial infection, overt HE grade or death) in hyperammonemic ACLF patients with no overt HE.

Study design:

* A Prospective Randomized Controlled Trial.
* Single Centre.
* Open label.
* Block Randomization will be done , it will be implemented by IWRS method.
* The study will be conducted in Department of Hepatology, ILBS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. ACLF as per APASL criteria (AARC grade I/II)
3. Baseline ammonia levels of ≥135ug/dl or 79.5umol/l
4. Given informed consent

Exclusion Criteria:

* 1. Overt HE 2. AARC grade III 3. Confirmed or suspected bacterial infection 4. Extrahepatic organ failure 5. Renal dysfunction lasting for more than 48 hours or need for vasoconstrictors 6. Paralytic ileus 7. Patients with hepatocellular carcinoma beyond Milan criteria or any other neoplastic disorder 8. Pregnant and lactating women 9. Use of lactulose, rifaximin or LOLA in past 48h 10. Uncontrolled DM, HT, CAD 11. Patients with allergy or other contraindications of the used drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving composite endpoint target NH3 level < 79.5 mmol/L (135mcg/dl) and /or Incidence of major adverse liver related outcomes (MALO) (any of AARC III, bacterial infection, overt HE grade or death) at day 7 in two arms. | Day 7

SECONDARY OUTCOMES:
Incidence of bacterial infection at day 4 and 7 in two arms | day 4 and 7
Incidence of overt HE at day 4 and 7 in two arms | day 4 and 7
Proportion of patients with AARC III ACLF at day 4 and 7 in two arms | day 4 and 7
Incidence of new AKI, SBP, Variceal bleed at day 4 and 7 in two arms | day 4 and 7
Proportion of patients with ammonia <79.5 mmol/L(135mcg/dl) at day 1,2,3 and day 7 in 2 arms | day 1,2,3 and day 7
Proportion of patients with >25% and 50% ammonia reduction at day 1,2,3 and day 7 in 2 arms | day 1,2,3 and day 7
Liver related mortality at day 28 and day 90 | day 28 and day 90
Changes in markers of systemic inflammation from baseline and day 7 in two arms | day 7
Adverse effect of ammonia lowering therapies | day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided